CLINICAL TRIAL: NCT01114919
Title: Helping Problem Drinkers on the Internet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Dr. John Cunningham, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 282/2009
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Alcohol Dependence
Keywords: Problem drinking; Alcohol dependence; Alcohol abuse; Internet based intervention; Treatment; Alcohol Use Disorders Identification Test
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Check Your Drinking (CYD) — Internet based program of lower intensity as compared to the "Alcohol Help Centre. It was designed to assesses drinking patterns, increase self-awareness of individual triggers, and set and achieve goals regarding abstinence.
Behavioral: Alcohol Help Centre (AHC) — Internet based program of higher intensity as compared to the "Check Your Drinking" intervention. It was designed to assesses drinking patterns, increase self-awareness of individual triggers, and set and achieve goals regarding abstinence.

SUMMARY:
The main aim of this study is to compare the impact of a minimal and a full Internet-based self-help intervention for problem drinkers in the general population.

DETAILED DESCRIPTION:
Many problem drinkers never access any treatment services. Because of the individual as well as societal costs of heavy alcohol consumption, it is essential to find ways to intervene and provide assistance to problem drinkers. The Internet takes treatment to problem drinkers rather than requiring them to come to treatment, resulting in increased options for help for alcohol abusers. There is a preponderance of internet websites which are designed for self change in areas that include alcohol use. To date, however, there has been minimal scientific evaluation regarding the efficacy and safety of such programs.

Our own previous research found that we could reduce alcohol consumption by about three drinks per week at a six-month follow-up using a minimal, personalized feedback Internet-based intervention. Building on this, the current project will attempt to increase the impact of Internet-based interventions as well as produce sustained reductions in drinking by adding an extended online self-help service to this already promising minimal intervention. More specifically, this randomized, double blinded study will compare and evaluate the efficacy of two different degrees of treatment intervention for problem drinkers: a minimal one ("Check your Drinking") and a full one ("Alcohol Help Centre").

ELIGIBILITY:
Inclusion Criteria:

* Resident of Ontario
* 19 years of age or over
* Have consumed alcohol in the one month prior to the telephone survey.
* Have consumed alcohol in the one month prior to the telephone survey.
* A score of 8 or over on the Alcohol Use Disorders Identification Test (AUDIT)
* Indicate an interest in receiving self-help materials
* Have home access to the Internet
* Are willing to participate in follow-up at six and twelve month intervals

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Frequency of consumption | 6 months and 12 months
Usual number of drinks per occasion | 6 months and 12 months
Frequency of consuming 5 or more drinks on one occasion | 6 months and 12 months
Typical weekly consumption | 6 months and 12 months
Highest number of drinks on one occasion | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cunningham JA. Comparison of two internet-based interventions for problem drinkers: randomized controlled trial. J Med Internet Res. 2012 Aug 1;14(4):e107. doi: 10.2196/jmir.2090. PMID 22954459
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre. — http://www.camh.net/research